CLINICAL TRIAL: NCT02522221
Title: A "Real-World", Randomized, Open-Label, Study on the Efficacy, Safety, and Tolerability of Tecarfarin (ATI-5923) a Novel Vitamin K Antagonist, Versus Warfarin in Subjects Requiring Chronic Anticoagulation
Brief Title: Tecarfarin Anti-Coagulation Trial (TACT)
Acronym: TACT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Espero Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-511
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Thromboembolism; Thrombosis
Keywords: chronic anticoagulation; vitamin K antagonist; mechanical heart valve; CYP2C9; warfarin; tecarfarin; chronic kidney disease
MeSH Terms: conditions — Thromboembolism; Thrombosis; Renal Insufficiency, Chronic | interventions — Warfarin; tecarfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tecarfarin (Experimental): Tecarfarin will be administered and dose adjusted by the investigator. Dose adjustments will be made in accordance with a target INR range pre-specified by the investigator.
  Interventions: Drug: tecarfarin
- Warfarin (Active Comparator): Warfarin will be administered and dose adjusted by the investigator. Dose adjustments will be made in accordance with a target INR range pre-specified by the investigator.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Warfarin is an oral vitamin K antagonist anticoagulant.
  Other Names: Coumadin
  Arms: Warfarin
Drug: tecarfarin — Tecarfarin is an oral vitamin K antagonist anticoagulant
  Other Names: ATI-5923
  Arms: Tecarfarin

SUMMARY:
TACT is a "real world" randomized controlled trial of tecarfarin, a novel vitamin K antagonist, vs. warfarin. The quality of anticoagulation control will be compared for the two groups of subjects who require chronic oral anticoagulation for a broad panel of indications.

DETAILED DESCRIPTION:
This will be a randomized, parallel-arm, open-label study comparing the safety and efficacy of tecarfarin and warfarin in approximately 1000 subjects who have an indication for chronic oral anticoagulation. The study will be fully enriched with subjects who are taking at least one CYP2C9-interacting medication and have either chronic kidney disease stage 3 or 4 and/or a genetic variant allele for CYP2C9. The study will be conducted at approximately 140 sites with experience in the management of anticoagulation subjects. Eligible subjects will be randomized to receive either tecarfarin or warfarin for a period ranging from 6 months to a maximum of approximately 24 months.

ELIGIBILITY:
General Screening Inclusion Criteria

1. Is male or female and at least 18 years of age.
2. Is able and willing to sign an IRB-approved written informed consent.
3. Is able and willing to follow instructions, to comply with protocol requirements, and to attend required study visits.
4. Is taking a CYP2C9-interacting medication (inhibitor, substrate, or inducer; see list in Appendix A) at the time of randomization and is expected to receive this medication chronically for the duration of the trial.
5. Has either

   1. Chronic kidney disease stage 3 or 4 (eGFR ≥ 15 to <60 mL/min/1.73 m2 at Screening based on central laboratory) and/or
   2. A CYP2C9 genotype variant allele
6. (Only for warfarin experienced patients) Patient is considered poorly controlled on warfarin therapy as judged by the investigator, e.g. has at least 2 INR values out of target range within previous 12 months Anticoagulation-Related Inclusion Criteria
7. Requires chronic anticoagulation therapy.
8. Is willing to receive chronic anticoagulation investigational therapy for the duration of the study or, for warfarin-naïve DVT subjects, treating physician prescribed at least a 6-month treatment period with an oral anticoagulation agent.
9. Has one or more of the following indications for chronic oral anticoagulation:

   1. Atrial fibrillation/flutter (paroxysmal, persistent or permanent), not due to a reversible cause, documented by electrocardiography (ECG)
   2. Aortic and/or mitral prosthetic HV
   3. History of venous thromboembolic disease
   4. History of myocardial infarction or cardiomyopathy
   5. Any another indication for which warfarin is approved or recommended, with Sponsor approval
10. Conforms to the following restrictions regarding vitamin-K containing dietary supplements:

    1. If taking at Baseline (Visit 2), is willing to continue with consistent doses throughout the study
    2. If not taking at Baseline (Visit 2), is willing to abstain from such supplements throughout the study

General Exclusion Criteria

1. Is pregnant, nursing, or a woman of childbearing potential who cannot assure that they will not become pregnant for the duration of the study.
2. Has been treated with an investigational drug within 30 days or 5 half-lives, whichever is longer, at time of screening.

   Safety-Related Exclusion Criteria
3. Has a life expectancy <1 year
4. Is age >85 years
5. Has severe end-organ disease, such as:

   1. Estimated GFR (eGFR) < 15 mL/min/1.73 m2 at Screening per the central laboratory
   2. Is on dialysis
   3. Is expected to be on dialysis or receive kidney transplant within 6 months of screening
   4. Advanced pulmonary disease requiring home oxygen
   5. NYHA class IV heart failure
   6. Severe psychiatric disorder such as advanced dementia
6. Has a history of ischemic stroke without residual neurologic deficit within the last 3 months, prior major ischemic stroke with residual neurologic deficit, or any history of intracranial bleeding
7. Is an ongoing alcohol or substance abuser
8. Has anemia (screening hemoglobin <9 g/dL) For subjects who have received a MHV within 4 weeks of Screening, who have no active bleeding, and whose hemoglobin is stable, a Screening hemoglobin as low as 8 g/dL is allowed.

   For subjects with severe CKD (eGFR ≥ 15 to <30 mL/min/1.73 m2), who have no active bleeding, and whose hemoglobin is stable, a Screening hemoglobin as low as 8 g/dL is allowed.
9. Has thrombocytopenia (screening platelet count <90,000 x 103/microL)
10. Has a history of or presence of any illness or condition, which, in the judgment of the Investigator, may compromise the safety of the subject during Study Drug administration.

    Anticoagulation-related Exclusion Criteria
11. Has active bleeding or lesions at risk of bleeding such as gastric ulceration, colonic or cerebral arterio-venous malformations, cerebral or aortic aneurysms, pericarditis or endocarditis
12. Except for MHV replacement surgery and related or concurrent procedures, has recently (<14 days from Screening) undergone non-thromboembolic surgery or other invasive procedures such as lumbar puncture.
13. Has blood dyscrasias or inherited disorders of hemostasis.
14. Has a history of hemorrhagic tendencies or prior serious hemorrhagic events such as hemorrhage within the cranium, eye, spinal cord, retroperitoneum.
15. Has active gross hematuria or gastrointestinal bleeding
16. Has a history of gross hematuria or gastrointestinal bleeding within the past 6 months prior to Screening. (Note: Investigators may enroll patients with such bleeding episodes if they are resolved at least 4 weeks prior to screening and if the benefits of anticoagulation outweigh the risks using accepted risk stratification methods such as HASBLED.)
17. Has received concomitant therapy with other anticoagulant or antiplatelet agents, such as clopidogrel, prasugrel, ticlopidine, dipyridamole, heparin or low molecular weight heparin (LMWH), or nonsteroidal anti-inflammatory drugs (NSAIDs) that cannot be discontinued prior to initiating tecarfarin/warfarin dosing, unless use of such drugs is necessary as part of bridging/transitioning during the first several days of Study Drug administration.

    Daily use of 81 - 100 mg aspirin and intermittent or chronic use of the selective COX-2 inhibitors celecoxib and valdecoxib is allowed.
18. Has congenital or acquired coagulant inhibitors present which would interfere with the use of the INR, eg:

    1. Antiphospholipid antibody syndrome or positive lupus anticoagulant
    2. Abnormally prolonged prothrombin time, in the absence of therapeutic anticoagulation, due to an endogenous inhibitor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in the therapeutic range (TTR) for tecarfarin vs. warfarin for each treatment group in the randomized population | From the date of randomization until study termination, up to 24 months (1st month not included)
  Interpolated and observed TTR will be calculated for the two treatment groups

SECONDARY OUTCOMES:
Percentage TTR for tecarfarin vs. warfarin in the sub-population of patients who are taking a CYP2C9-interacting medication and have a CYP2C9 genotype variant allele | From the date of randomization until study termination, up to 24 months (1st month not included)
  Interpolated and observed TTR will be calculated for the two treatment groups
Percentage TTR for tecarfarin vs warfarin for the sub-population of patients who are taking a CYP2C9-interacting medication and have chronic kidney disease stage 3 or 4 (eGFR ≥ 15 to <60 mL/min/1.73 m2) | From the date of randomization until study termination, up to 24 months (1st month not included)
  Interpolated and observed TTR will be calculated for the two treatment groups
Percentage of patients with INR > 4.0 for tecarfarin vs. warfarin | From the date of randomization until study termination, up to 24 months (1st month not included)
  Percentage of observations of patients with INR > 4.0 will be calculated for the two treatment groups
Percentage of patients with INR > 5.0 | From the date of randomization until study termination, up to 24 months (1st month not included)
  Percentage of observations of patients with INR > 5.0 will be calculated for the two treatment groups
Time to first embolic event for tecarfarin vs. warfarin | From the date of randomization until study termination, up to 24 months
  Time from enrollment until any embolic event (CVA, pulmonary embolism, peripheral embolism) while enrolled will be calculated for the two groups

OTHER OUTCOMES:
The primary safety endpoint of this study is the time to the first BARC category 3-5 bleeding event. | From the date of randomization until study termination, up to 24 months
  BARC category 3-5 bleeding events will be compared for the two treatment groups
The secondary safety endpoint of this study is the time to the first BARC category 2-5 bleeding event | From the date of randomization until study termination, up to 24 months
  BARC category 2-5 bleeding events will be compared for the two treatment groups